CLINICAL TRIAL: NCT06513585
Title: The First Affiliated Hospital of Xinjiang Medical University
Brief Title: Primary Aldosteronism: Superselective Embolization vs. Laparoscopic Endocrine Curative Therapy
Acronym: PA-SELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinjiang Medical University (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Head of Hypertension Department, Clinical Professor, Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240613
Record Dates: First submitted 2024-06-24; First posted 2024-07-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Primary Aldosteronism; Suprarenalectomy; Super Selective Adrenal Artery Embolization
MeSH Terms: conditions — Hyperaldosteronism | interventions — Adrenalectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superselective adrenal artery embolization group (Experimental): Superselective adrenal artery embolization for primary aldosteronism
  Interventions: Procedure: Superselective adrenal artery embolization or adrenalectomy
- Adrenalectomy group (Active Comparator): Adrenalectomy for primary aldosteronism
  Interventions: Procedure: Superselective adrenal artery embolization or adrenalectomy

INTERVENTIONS:
Procedure: Superselective adrenal artery embolization or adrenalectomy — Arm A underwent SAAE treatment, and arm B underwent laparoscopic adrenalectomy.
  Other Names: Adrenalectomy

SUMMARY:
The aim of this study was to compare the efficacy and safety of adrenalectomy and superselective adrenal artery embolization in a prospective, multicenter, randomized controlled study. To provide a new interventional alternative therapy for primary aldosteronism.

DETAILED DESCRIPTION:
Primary hyperaldosteronism is caused by excessive aldosterone secretion caused by adrenal cortex disease, which leads to increased sodium and potassium discharge, increased fluid volume and inhibition of renin-angiotensin-aldosterone system. It is one of the common causes of secondary hypertension as clinical symptoms with hypertension, hypokalemia, hyperaldosterone and low renin. It accounts for 5% to 13% of people with hypertension. In addition to the impact of hypertension itself on the body, the endocrine hormone disorder and electrolyte imbalance associated with PA may also become independent risk factors for cardiovascular and cerebrovascular events, and the risk of stroke, atrial fibrillation and myocardial infarction is significantly higher than that of essential hypertension, so early detection and reasonable treatment are crucial. PA can be divided into 6 types according to the etiology, of which the most common is idiopathic aldosteronism (IHA) and aldosteronoma, accounting for 60% and 30% respectively, unilateral adrenal hyperplasia followed, the other subtypes are less common. Previous guidelines have recommended surgery and drug intervention as the main measures for the treatment of PA, while unilateral PA is preferred by surgery and laparoscopic adrenalectomy. However, surgical treatment also has many limitations: First, not all patients with surgical indications have the opportunity to undergo adrenal resection. Surgical treatment is not suitable for patients with difficult laparoscopic operation, such as obesity, serious abdominal adhesion due to previous surgical history, and high-risk surgery, such as cardiovascular and cerebrovascular diseases and emphysema. In addition, adrenal resection may lead to adrenal dysfunction, serious infection, retroperitoneal hematoma and many other adverse reactions. The efficacy and safety of superselective adrenal artery embolization as a new alternative therapy for PA intervention have been proved. The aim of this study was to compare the efficacy of adrenectomy and superselective adrenal artery embolization according to international PASO evaluation criteria, and to conduct a prospective, multicenter, randomized controlled study in Xinjiang to explore the potential of SAAE as a treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Diagnosed with primary aldosteronism according to the 2016 Clinical guidelines of the International Endocrine Society
* Primary aldosteronism diagnosed according to international guidelines Unilateral disease by AVS or PET-CT criteria
* Patients and their family members signed informed consent and agreed to participate in the study

Exclusion Criteria:

* A history of severe hypersensitivity to contrast media
* Severe liver disease complications, such as thrombocytopenia, esophageal varices rupture bleeding, etc
* Renal insufficiency (serum creatinine > 176mmol/L or estimated glomerular filtration rate < min.1.73m2)
* Combined with other secondary hypertension, such as pheochromocytoma, hypercortisolism, renal vascular hypertension (such as renal artery stenosis), renin secretory tumor, renal parenchymatous hypertension, drug-induced hypertension (such as long-term use of glucocorticoids, contraceptives, estrogen, herbal medicines containing glycyrrhizin), pregnancy hypertension and other secondary hypertension
* Combined with genetic diseases: such as false aldosteronism (Liddle syndrome), Bartter syndrome, familial hypokalemia and hypomagnesia (Gitelman syndrome)
* Stroke, myocardial infarction and stent implantation occurred in the past 3 months
* Serious other diseases, such as heart dysfunction (grade IV), acute infections, autoimmune diseases, various malignant tumors, etc
* Participated in other clinical trials within the past 3 months
* Pregnant, breastfeeding, or planning a pregnancy
* Identify patients with alcohol allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete biochemical cure of PA | 6 months post intervention
  Complete biochemical cure of PA, defined (whilst off medications that might alter serum potassium or the RAS) by both:
  Normalisation of serum potassium, and Normalisation of ARR, or Elevated ARR and i). Baseline PAC <190pmol/L, or ii). Normal confirmatory test (as defined in the inclusion criteria)
Complete clinical cure of PA | 6 months post intervention
  Complete clinical cure of PA, defined as normotension without antihypertensive medication

SECONDARY OUTCOMES:
Changes in ambulatory blood pressure and baseline blood pressure | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  24-hour ambulatory blood pressure and office systolic and diastolic pressure
Change of the number of antihypertensive medications | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of the number of antihypertensive medications
Adverse events | Reported throughout the study period. Approximately 2 years
  Will be directly sought at each study visit through history and physical examination where appropriate Subjects will be encouraged to report between study visits and will have a mechanism to do so Will be classified by system, seriousness, causal relationship and expectedness according to the Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Readmission rate | Reported throughout the study period. Approximately 2 years
  Readmission rate, defined as readmission for primary aldosteronism
Change of blood electrolytes (K+, Na +) | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of blood electrolytes (K+, Na + in mmol/L)
Change of plasma aldosterone | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of plasma aldosterone (pg/mL)
Change of plasma cortisol | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of plasma cortisol (nmol/L)
Change of plasma renin measured | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of plasma renin (pg/ml)
Change of liver enzymes | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of liver enzymes (ALT, AST in IU/L)
Change of kidney function | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of serum creatinine in umol/L
Change of fasting blood glucose | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of fasting blood glucose in mmol/L
Change of lipids profiles | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L
Change of 24-h urine microalbumin | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of 24-h urine microalbumin (mg/L)
Change of 24-h 24-h urine creatinine | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of 24-h urine creatinine (umol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Ying Zheng, PhD, Study Chair — 1st affiliatted hospital of Xinjiang Medical University
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No